CLINICAL TRIAL: NCT03980743
Title: Adaptation of an Evidence-based Interactive Obesity Treatment Approach (iOTA) for Obesity Prevention in Early Serious Mental Illness: iOTA-eSMI
Brief Title: Interactive Obesity Treatment Approach for Obesity Prevention in Adults With Early Serious Mental Illness: iOTA-SMI
Acronym: iOTA-eSMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201911123
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Overweight; Severe Mental Disorder
Keywords: Obesity; Overweight; Severe Mental illness
MeSH Terms: conditions — Obesity; Overweight; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iOTA text messaging intervention (Active Comparator): There will be a 6 month "active" treatment phase consisting of monthly meetings with a study health coach to develop reasonable health goals and interactive text messaging to provide daily support and self-monitoring of behavior change goals between in-person visits. Participants may receive phone calls between visits from their health coach for additional support if needed. Following the active treatment phase, participants will receive daily health-related text messages for another 3 months.
  Interventions: Behavioral: iOTA text messaging intervention
- Health Education text messaging intervention (Placebo Comparator): There will be a 6 month "active" treatment phase consisting of monthly in-person visits with a health coach to learn about healthy eating and activity behaviors, including developing readiness for health behavior change. Participants will not set specific health goals, but will receive weekly text messages about general health tips related to their in-person visits. Following the active treatment phase, participants will receive daily health-related text messages for another 3 months.
  Interventions: Behavioral: Health Education text messaging intervention

INTERVENTIONS:
Behavioral: iOTA text messaging intervention — Over 6 months, participants in the iOTA arm will have monthly in-person visits with a health coach who will work with the participant to set goals for the upcoming month related to healthy eating and activity. The participant will receive daily text message health tips related to their goals, and will be prompted once a week to respond with a text indicating their weight and how they are doing with their goals. Following the 6-month active treatment phase, participants will receive text messages only for another 3 months.
  Other Names: iOTA
  Arms: iOTA text messaging intervention
Behavioral: Health Education text messaging intervention — Over 6 months, participants in the Health Ed arm will also have monthly in-person visits with a health coach who will provide education on energy balance and problem-solving. Specific goals will not be set, but the health coach will assist participants in problem-solving any challenges. Participants will receive a weekly automated motivational text message health tip from the study related to what they learned in their health coaching sessions. Following the 6-month active treatment phase, participants will receive text messages only for another 3 months.
  Other Names: Health Ed
  Arms: Health Education text messaging intervention

SUMMARY:
Using a design-for-dissemination approach, this application proposes to use combined methods to adapt and pilot test an interactive obesity treatment approach (iOTA) for obesity prevention in early serious mental illness (eSMI) that uses text messaging to provide between-visit support. Derived from the lifestyle intervention used in the Diabetes Prevention Program, the parent iOTA targets diet, activity and adherence using web-based and health coach support.

DETAILED DESCRIPTION:
Most obesity and related complications in serious mental illness (SMI) occur in the context of chronic psychiatric illness, but there are few treatments that work. Behavioral interventions face challenges with long-term effectiveness, implementation and sustainability. Medications have modest effectiveness at best, and/or pose serious side effect risks. This study focuses on prevention of chronic obesity by adapting and pilot testing a prevention-focused, interactive obesity treatment approach (iOTA) for use in persons with early-phase SMI (eSMI) experiencing initial weight gain, overweight or early-stage obesity. The intervention will be adapted from the most studied, effective iOTA, derived from the Diabetes Prevention Program. The parent iOTA uses health coaches who extend their sustainable reach with scalable, inexpensive, semi-automated text messaging. Using a formal evaluation process and a specific implementation science framework, planned adaptations for this application will address mechanisms to improve health-related awareness, insight and self-efficacy skills.

Aim 1: Evaluate barriers and facilitators for intervention engagement, effectiveness and implementation, and identify needed adaptations of the prior iOTA for use in obesity attenuation in eSMI.

Aim 2: Adapt the prior iOTA for use in obesity attenuation in eSMI, aiming to maximize acceptability, engagement, sustainable reach and target engagement for eSMI.

Aim 3: Conduct a randomized pilot and feasibility study of iOTA-eSMI in a diverse sample of adults aged 18-45 with eSMI and initial weight gain, overweight or early class I obesity, comparing iOTA-eSMI to a health education condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* At-risk weight defined as greater than 7 percent weight gain in the prior 2 years, overweight as evidenced by BMI 25-29.9, OR class I obesity as evidenced by BMI 30-32.49
* Serious Mental Illness diagnosis
* Receiving case management services
* University of California, San Diego Brief Assessment of Capacity to Consent score less than 14
* Not taking weight loss medications or participating in another behavioral weight loss intervention
* Mild to moderate psychiatric symptom severity as measured by the Clinical Global Impression Severity scale
* Willing and able to provide written informed consent

Exclusion criteria:

* Taking weight loss medications or participating in another behavioral weight loss intervention
* University of California, San Diego Brief Assessment of Capacity to Consent score greater than or equal to 14
* Acute suicidality at time of screening
* Unwilling or unable to provide written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ginger Nicol, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - South Florida Behavioral Health Network, Miami, Florida
  - Washington University in St. Louis Medical School, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicol GE, Jansen MO, Ricchio AR, Schweiger JA, Keenoy KE, Miller JP, Morrato EH, Guo Z, Evanoff BA, Parks JJ, Newcomer JW. Adaptation of a Mobile Interactive Obesity Treatment Approach for Early Severe Mental Illness: Protocol for a Mixed Methods Implementation and Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Jun 9;12:e42114. doi: 10.2196/42114. PMID 37294604

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | iOTA Text Messaging Intervention | Health Education Text Messaging Intervention
Started | 33 | 17
Completed | 18 | 9
Not Completed | 15 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iOTA Text Messaging Intervention | Health Education Text Messaging Intervention | Total
Number analyzed (Participants) | 33 | 17 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 17 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (11.2) | 39.8 (11.6) | 37.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 16 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 3 | 12
  Not Hispanic or Latino | 21 | 12 | 33
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 9 | 24
  White | 12 | 5 | 17
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 17 | 50
Marital Status [Count of Participants; unit: Participants]
  Single | 29 | 11 | 40
  Married/common law | 1 | 2 | 3
  Divorced | 2 | 1 | 3
  Unknown or not reported | 1 | 3 | 4
Employment [Count of Participants; unit: Participants]
  Employed | 4 | 3 | 7
  Unemployed | 22 | 10 | 32
  Unknown | 7 | 4 | 11
Income [Count of Participants; unit: Participants]
  0-$25,000 | 27 | 10 | 37
  $25,000 - 50,000 | 4 | 2 | 6
  >= $100,000 | 0 | 1 | 1
  Unknown or not reported | 2 | 4 | 6
Device Type [Count of Participants; unit: Participants]
  Smartphone | 32 | 16 | 48
  Unknown or not reported | 1 | 1 | 2
Insurance [Count of Participants; unit: Participants]
  Medicaid | 22 | 9 | 31
  Medicare | 3 | 3 | 6
  Commercial | 3 | 4 | 7
  Unknown or not reported | 5 | 1 | 6
Primary Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia Spectrum | 18 | 5 | 23
  Bipolar Mood Disorder | 6 | 5 | 11
  Major Depressive Disorder | 2 | 4 | 6
  Anxiety | 1 | 0 | 1
  PTSD | 3 | 2 | 5
  Autism | 1 | 0 | 1
  Unknown or not reported | 2 | 1 | 3
Weight (kg) [Mean (Standard Deviation); unit: Kilogram] | 110.1 (31.0) | 119.8 (34.0) | 113.5 (32.0)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 43.1 (11.5) | 38.1 (10.5) | 39.8 (11.0)
9-item Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire is a 9-item scale that assessed overall depression. A total score is reported with a range of 0 to 27, where a higher score represents worse overall depression. Population: Six participants withdrew their consent, and there was 1 participant missed the baseline session.
  A total number of 43 participants had the measures.
  units on a scale
    number analyzed (Participants) | 28 | 15 | 43
    (all) | 6.18 (6.40) | 7.73 (8.36) | 6.72 (7.09)
Self-efficacy for Diet & Exercise [Mean (Standard Deviation); unit: units on a scale] — This measure consists of 32 questions that assess over eating and exercise habits. Within it, there are 20 questions about the eating habits sub-scale and 12 questions about the exercise habits sub-scale. A total score is reported with a range of 32 to 160, where a lower score represents worse overall eating and exercise habits. Population: 6 participants withdrew consents, and 2 participants missed the baseline session
  units on a scale
    number analyzed (Participants) | 27 | 15 | 42
    (all) | 116.67 (29.53) | 124.27 (19.31) | 119.38 (26.34)
Loss of Control Over Eating Scale (LOCES) [Mean (Standard Deviation); unit: units on a scale] — Population: Six participants withdrew their consent, and there was 1 participant missed the baseline session.
  A total number of 43 participants had the measures.
  units on a scale
    number analyzed (Participants) | 28 | 15 | 43
    (all) | 15.1 (8.2) | 15.9 (7.8) | 15.4 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index
Description: weight in kilograms/height in meters squared
Time Frame: baseline and 24 weeks
Population: All participants have baseline measurements; only 18 iOTA participants and 9 participants in the Education group completed the 24-week follow-up.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | iOTA Text Messaging Intervention | Health Education Text Messaging Intervention
Number analyzed (Participants) | 33 | 17
kg/m^2
  baseline | 43.1 (11.5) | 38.1 (10.5)
  week24_endpoint: number analyzed (Participants) | 18 | 9
  week24_endpoint | 40.3 (13.3) | 40.3 (9.3)
Statistical Analysis 1: Comparison: iOTA Text Messaging Intervention vs Health Education Text Messaging Intervention; Time x treatment (week 0 and week 24); Test type: Superiority; p = 0.97, Mixed Models Analysis

2. Secondary Outcome: Change in Self-Efficacy for Diet and Exercise
Description: This questionnaire includes 32 questions in two domains of self efficacy: 1) healthy eating and 2) exercise.
  Within it, there are 20 questions about the eating habits sub-scale and 12 questions about the exercise habits sub-scale.
  Respondents are asked to recall how confident they have felt in doing positive health behaviors since the last study visit.
  Responses are on a likert scale of 1 - 5 (1 - 2 = I know I cannot do; 3 - 4 = Maybe I can; 5 = I know I can).
  A total score is reported with a range of 32 to 160, where a lower score represents worse overall eating and exercise habits.
  Total scores is measured at baseline and 24 weeks follow-up.
Time Frame: Baseline and 24 weeks
Population: One patient missed/ skipped this session in iOTA group at baseline; Only 7 participants in Education group and 9 iOTA participant completed the 24 weeks follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Education Text Messaging Intervention | iOTA Text Messaging Intervention
Number analyzed (Participants) | 15 | 28
score on a scale
  baseline: number analyzed (Participants) | 15 | 27
  baseline | 124.27 (4.99) | 116.67 (5.68)
  24 weeks: number analyzed (Participants) | 7 | 9
  24 weeks | 131.71 (9.45) | 109.67 (11.82)
Statistical Analysis 1: Comparison: Health Education Text Messaging Intervention vs iOTA Text Messaging Intervention; Time x treatment (week 0 and week 24) for Healthy Eating; Test type: Superiority; p = 0.273, Mixed Models Analysis

3. Secondary Outcome: Change in Psychophysical Skills & Insight
Description: This questionnaire includes 10 questions, with three separate subscales: 1)Self-determination, 2)Cognitive control and 3)Interoceptive Awareness).
  Respondents are asked to rate their own skills since the last study visit. Responses are on a likert scale of 1-5 (1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always).
  Scores are generated for each subscale, as well as a total score. Total score is from 10-50.
  Higher scores indicate greater degree of psychophysical awareness & skills.
Time Frame: Baseline and 24 weeks
Population: Time X treatment (0 and 24 weeks) with sum of the score
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Education Text Messaging Intervention | iOTA Text Messaging Intervention
Number analyzed (Participants) | 15 | 28
score on a scale
  baseline | 34.93 (1.56) | 33.36 (1.02)
  24 weeks: number analyzed (Participants) | 7 | 8
  24 weeks | 38.43 (2.20) | 35.50 (2.31)
Statistical Analysis 1: Comparison: Health Education Text Messaging Intervention vs iOTA Text Messaging Intervention; Test type: Superiority — Time x treatment (week 0 and week 24) with sum score; p = 0.691, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: The time frame is until the study's completion, an average of 6 months.
Description: No AEs/SAEs occurred through the study completion.
Arm/Group | iOTA Text Messaging Intervention | Health Education Text Messaging Intervention
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/17
Other Adverse Events (participants affected / at risk) | 0/33 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT03980743/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT03980743/SAP_001.pdf
  • Informed Consent Form (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT03980743/ICF_002.pdf